CLINICAL TRIAL: NCT01168791
Title: A Phase III Multicenter, International, Randomized, Double-blind, Placebo-controlled Study of Doxorubicin Plus Palifosfamide-tris vs. Doxorubicin Plus Placebo in Patients With Front-line Metastatic Soft Tissue Sarcoma.
Brief Title: Study of Palifosfamide-tris in Combination With Doxorubicin in Patients With Front-line Metastatic Soft Tissue Sarcoma
Acronym: PICASSO III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IPM3001
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Soft Tissue Sarcoma
Keywords: Metastatic; Front line
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis | interventions — Doxorubicin; isophosphamide mustard

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- doxorubicin plus palifosfamide-tris (Experimental)
  Interventions: Drug: doxorubicin in combination with palifosfamide-tris
- doxorubicin plus placebo (Active Comparator)
  Interventions: Drug: doxorubicin in combination with placebo

INTERVENTIONS:
Drug: doxorubicin in combination with palifosfamide-tris — palifosfamide-tris: 150 mg/m2 3 days every 21 days for a maximum of 6 cycles.
  doxorubicin: 75 mg/m2 1 day every 21 days for a maximum of 6 cycles.
  Arms: doxorubicin plus palifosfamide-tris
Drug: doxorubicin in combination with placebo — doxorubicin: 75 mg/m2 of doxorubicin 1 day every 21 days for a maximum of 6 cycles.
  placebo: 250 mL of normal saline 3 days every 21 days for a maximum of 6 cycles.
  Arms: doxorubicin plus placebo

SUMMARY:
This is an international, randomized, double-blind, placebo-controlled trial to evaluate the clinical efficacy of palifosfamide-tris administered with doxorubicin in combination, compared with doxorubicin administered with placebo in front-line patients diagnosed with metastatic soft tissue sarcoma (STS).

ELIGIBILITY:
To be eligible, each patient must meet EACH of the following criteria:

* Age ≥18 years.
* Documented soft tissue sarcoma
* Metastatic disease for which the patient has not received any prior treatment, and for whom treatment with doxorubicin is considered medically acceptable.
* ECOG Performance Status of 0, 1 or 2
* Adequate bone marrow and organ function based on the results of protocol- specified laboratory tests
* Male and female patients must agree to use a highly reliable method of birth control during study participation.
* Able to provide informed consent

To be eligible, each patient must meet NONE of the following criteria:

* Specific sarcoma histological subtypes including GIST and Ewing's sarcoma.
* Systemic therapy for the treatment of metastatic sarcoma, prior to or during the study. However, patients may have received neo-adjuvant/adjuvant Gemzar and Taxotere chemotherapy for their primary sarcoma, prior to the development of metastatic disease
* Any prior anthracycline use.
* Known allergy to any of the study drugs or their excipients.
* Any unstable or clinically significant concurrent medical condition that would, in the opinion of the investigator, jeopardize the safety of a patient and/or their compliance with the protocol, based on screening tests, physical examination and medical history (as specifically defined in the clinical protocol).
* Myocardial dysfunction defined as left ventricular ejection fraction (LVEF) <50%.
* Documented metastases to brain or meninges.
* Any malignancy other than sarcoma within the last 5 years prior to screening, with the exception of cervical carcinoma in situ, basal cell carcinoma, or superficial bladder tumors (Ta, Tis, or T1) that have been successfully and curatively treated with no evidence of recurrent or residual disease.
* Currently pregnant or nursing.
* Radiotherapy with curative intent within 4 weeks of first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2010-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival followed by Overall Survival | assessed every 6 weeks for 22 weeks, then 8 weeks for 6 months/until progression, then every 12 weeks until then death

SECONDARY OUTCOMES:
Quality of Life, as assessed by EORTC QLQ-C30 and EQ-5D questionnaires | assessed every 6 weeks for 22 weeks, then 8 weeks for 6 months, then every 12 weeks until death
Safety and Tolerability as evaluated using CTCAE v 4.0 | 22 weeks

CONTACTS AND LOCATIONS:
Locations (161):
- United States (73):
  - Birmingham, Alabama
  - Arizona Oncology Associates, Phoenix, Arizona
  - Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California, Los Angeles, Los Angeles, California
  - Los Angeles, California
  - University of California, Irvine, Orange, California
  - Pomona, California
  - Sarcoma Oncology Center, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Medical Oncology Hematology Consultants, Newark, Delaware
  - MedStar Research Institute, Washington D.C., District of Columbia
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Emory, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Kootenai Cancer Center, Post Falls, Idaho
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Indiana University Simon Cancer Center, Indiannapolis, Indiana
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Kansas City Cancer Center, Overland Park, Kansas
  - New Orleans, Louisiana
  - LSU Health Sciences Center, Feist-Weiller Cancer Center, Shreveport, Louisiana
  - Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St.Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Las Vegas, Nevada
  - Hackensack, New Jersey
  - Morristown, New Jersey
  - Saint Barnabas, West Orange, New Jersey
  - Albuquerque, New Mexico
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - UC Cancer Institute, Cinncinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Cancer Care Associates, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Bethelehem, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Oncology/Hematology Associates, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Texas Oncology, Bedford, Texas
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Burlington, Vermont
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington
  - Bellin Cancer Center, Green Bay, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
  - Milwaukee, Wisconsin
- Argentina (5):
  - Ciudad de Buenos Aires
  - Córdoba
  - Ramos Mejía
  - Instituto CAICI, Rosario
  - Sante Fe
- Australia (10):
  - North Adelaide Oncology, Adelaide
  - Royal Adelaide Hospital, Adelaide
  - Camperdown
  - East Melbourne
  - The Canberra Hospital, Garran
  - Garran
  - Kurralta Park
  - Nedlands
  - Prince of Wales Hospital, Randwick
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (4):
  - Antwerp
  - Brussels
  - Leuven
  - Liège
- Brazil (10):
  - Institution name: Hospital de Câncer de Barretos - Fundação PIOXII, Barretos
  - Belo Horizonte
  - Santa Casa da Misericórdia de Curitiba, Curitiba
  - Florianópolis
  - Jaú
  - Hospital da Cidade de Passo Fundo, Passo Fundo
  - Hospital das Clínicas de Porto Alegre, Porto Alegre
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Centro de Oncologia da Bahia, Salvador
  - São Paulo
- Canada (5):
  - Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Mount Sinai Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University, Montreal, Quebec
- Chile (3):
  - Santiago
  - Instituto Clínico Oncológico del Sur, Temuco
  - Viña del Mar
- Colombia (3):
  - Bogotá
  - Medellín
  - Montería
- France (9):
  - Angers
  - Bordeaux
  - Institut Paoli Calmettes, Marseille
  - Marseille
  - Montpellier
  - Nice
  - Paris
  - Toulouse
  - Villejuif
- Germany (5):
  - HELIOS Klinikum Berlin Buch, Bad Sarrow
  - Universitätsklinikum Köln, Cologne
  - Hanover
  - Mannheim
  - Tuebingen University Hospital, Tübingen
- Guatemala City, Guatemala
- India (5):
  - Jaipur
  - Mumbai
  - Nashik
  - Pune
  - Secunderabad
- Israel (6):
  - Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Italy (3):
  - Candiolo
  - Humanitas Cancer Center, Rozzana
  - Ospedale Gradenigo Oncology, Torino
- Panama (2):
  - Centro Hemato Oncologico Paitilla, Panama City
  - Medical and Research Center, Panama City
- Poland (3):
  - Wojewodzkie Centrum Onkologii, Gdansk
  - Gilwice
  - Centrum Onkologii Instytut, Warsaw
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Craiova
- Russia (4):
  - Moscow
  - Obninsk
  - Saint Petersburg
  - Yaroslavl
- Singapore, Singapore
- Spain (4):
  - Badalona
  - Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Valencia
- United Kingdom (2):
  - The Royal Marsden NHS Foundation Trust Sarcoma, London
  - Christie Hospital NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Ryan CW, Merimsky O, Agulnik M, Blay JY, Schuetze SM, Van Tine BA, Jones RL, Elias AD, Choy E, Alcindor T, Keedy VL, Reed DR, Taub RN, Italiano A, Garcia Del Muro X, Judson IR, Buck JY, Lebel F, Lewis JJ, Maki RG, Schoffski P. PICASSO III: A Phase III, Placebo-Controlled Study of Doxorubicin With or Without Palifosfamide in Patients With Metastatic Soft Tissue Sarcoma. J Clin Oncol. 2016 Nov 10;34(32):3898-3905. doi: 10.1200/JCO.2016.67.6684. Epub 2016 Sep 30. PMID 27621408